CLINICAL TRIAL: NCT02277431
Title: A Randomized Controlled Trial of a Commercially-Available Probiotic Supplement (Trenev Trio®/Healthy Trinity®) and the Promotion of Normal Gastrointestinal Function Among Adults With Recurrent Gastrointestinal Symptoms
Brief Title: Probiotic Supplementation Among Adults With Recurrent Gastrointestinal Symptoms
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Chris D'Adamo, Assistant Professor Department of Family and Community Medicine Department of Epidemiology and Public Health Director of Research Center for Integrative Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 00007145
Record Dates: First submitted 2014-10-24; First posted 2014-10-29 (Estimated); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Gastrointestinal Symptoms; Bloating; Gas; Indigestion; Abdominal Pain; Defecation Irregularity
MeSH Terms: conditions — Mucopolysaccharidosis IV; Dyspepsia; Abdominal Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic dietary supplement (Experimental): Trenev Trio® (healthcare professional line)/Healthy Trinity® (consumer line) is a dietary supplement that contains probiotics microenrobed in an oil matrix in a two-piece hard gel capsule. One capsule will be taken twice per day (am & pm) offering a total daily serving of:
  * Lactobacillus acidophilus NAS super strain (10 billion Colony Forming Units [CFU])
  * Bifidobacterium bifidum Malyoth super strain (40 billion CFU)
  * Lactobacillus delbrueckii subspecies bulgaricus LB-51 super strain (10 billion CFU)
  Interventions: Dietary Supplement: Probiotic dietary supplement (Trenev Trio®)
- Placebo (Placebo Comparator): The placebo capsules utilized in this study will be indistinguishable from the probiotic dietary supplement capsules as they will be identical in appearance, odor, weight, and taste. Furthermore, the same sunflower oil matrix will be in both the probiotic dietary supplement and placebo. The only difference between the dietary supplement and placebo capsules will be the probiotic bacteria.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Probiotic dietary supplement (Trenev Trio®) — Trenev Trio® (healthcare professional line)/Healthy Trinity® (consumer line) is a dietary supplement that contains probiotics microenrobed in an oil matrix in a two-piece hard gel capsule. One capsule will be taken twice per day (am & pm) offering a total daily serving of:
  * Lactobacillus acidophilus NAS super strain (10 billion Colony Forming Units [CFU])
  * Bifidobacterium bifidum Malyoth super strain (40 billion CFU)
  * Lactobacillus delbrueckii subspecies bulgaricus LB-51 super strain (10 billion CFU)
  Arms: Probiotic dietary supplement
Dietary Supplement: placebo
  Arms: Placebo

SUMMARY:
Participants experiencing recurrent gastrointestinal symptoms in this double-blind, randomized, controlled trial will receive either a commercially-available probiotic dietary supplement or placebo. The investigators hypothesize that participants in the probiotic dietary supplement group will experience greater improvement in their gastrointestinal symptoms than participants in the placebo group.

ELIGIBILITY:
Inclusion Criteria:

1. Self-reported response of "moderate discomfort" or worse (3 or greater on 1-5 Likert Scale) and "frequent discomfort" or more often (3 or greater on 1-5 Likert scale) from at least 2 of the following gastrointestinal symptoms: gas, indigestion, bloating, abdominal pain, or defecation irregularity as expressed on Likert scale (1=very minor or no discomfort, 2=minor discomfort, 3=moderate discomfort, 4=high discomfort, 5=very high discomfort) over the previous 3 weeks
2. Agree to continue with typical diet and exercise habits during study
3. Agree to use contraception or abstinence throughout study period, unless postmenopausal or surgically sterile (females only)
4. Able to understand and voluntarily consent to the study and understand its nature and purpose including potential risks and side effects

Exclusion Criteria:

1. Current and documented diagnosis of Inflammatory Bowel Disease (Crohn's disease or ulcerative colitis), Celiac disease, active peptic ulcer, active diverticulitis, and other active cases of gastrointestinal diseases that, in the investigators' opinions, may affect participant safety.
2. Current and documented diagnosis of any other non-gastrointestinal disease that, in the investigators' opinions, may affect participant safety or confound the evaluation of the study outcomes. Excluded conditions include congestive heart failure, malignancy, uncontrolled diabetes mellitus, uncontrolled autoimmune disease (lupus, rheumatoid arthritis, eczema), eating disorders, and any other active health condition or disease that the investigators feel contradict the intended study population of participants in good health.
3. Daily consumption of another probiotic supplement or new consumption of fermented dairy products (yogurt, kefir, etc.)
4. Usage of systemic steroids during the past 2 months
5. Usage of antipsychotic medications during the past 2 months
6. Usage of prednisone, 6-mercaptopurine, adalimumab, etanercept, infliximab, leflunomide, golimumab, or mycophenolate mofetil during the past 2 months
7. Uncontrolled anxiety or current medication for anxiety disorder
8. Pregnant or breastfeeding females
9. History of alcohol, drug, or medication abuse
10. Known allergies to any substance in the study product
11. Previous major gastrointestinal tract surgery (colon resection, gastric bypass, etc.)
12. Participation in another clinical trial within 30 days of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-12; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Severity of self-reported bloating | Study end (6 weeks from baseline)
  Likert scale
Severity of self-reported gas | Study end (6 weeks from baseline)
  Likert scale
Severity of self-reported indigestion | Study end (6 weeks from baseline)
  Likert scale
Severity of self-reported abdominal pain | Study end (6 weeks from baseline)
  Likert scale
Severity of self-reported defecation irregularity | Study end (6 weeks from baseline)
  Likert scale

SECONDARY OUTCOMES:
Frequency of self-reported bloating | Study end (6 weeks from baseline)
  Likert scale
Frequency of self-reported gas | Study end (6 weeks from baseline)
  Likert scale
Frequency of self-reported indigestion | Study end (6 weeks from baseline)
  Likert scale
Frequency of self-reported abdominal pain | Study end (6 weeks from baseline)
  Likert scale
Frequency of self-reported defecation irregularity | Study end (6 weeks from baseline)
  Likert scale

OTHER OUTCOMES:
Gastrointestinal Symptom Rating Scale | Study end (6 weeks from baseline)
Gastrointestinal Quality of Life Index | Study end (6 weeks from baseline)
Bristol Stool Scale | Study end (6 weeks from baseline)
Rescue medication usage | Study end (6 weeks from baseline)
Adequate relief | Study end (6 weeks from baseline)
  "In the past 7 days, have you had adequate relief of your gastrointestinal discomfort?"

CONTACTS AND LOCATIONS:
Overall Officials: Chris D'Adamo, PhD, Principal Investigator — University of Maryland, College Park